CLINICAL TRIAL: NCT00668681
Title: Safety Data Collection for Delivery System and Use of Staple in Endovascular Procedures
Brief Title: Evaluation of EndoRefix Endovascular Delivery System and Staple
Acronym: EndoRefix
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company business decision, IDE closed, no commercialization planned
Sponsor: Lombard Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endo060234
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: AAA Graft Implant for Primary Aneurysm Treatment; AAA Graft Repair to Extend Life of Implant
Keywords: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endorefix (Active Comparator): Evaluation of EndoRefix Endovascular Delivery System and Staple
  Interventions: Device: EndoRefix

INTERVENTIONS:
Device: EndoRefix

SUMMARY:
This study is intended to provide data to verify safe delivery of a staple previously intended for use in open surgical procedures. A newly modified delivery system will provide endovascular access for implantation of a staple during endovascular graft procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >21 years of age
2. Undergoing endovascular stent grafting for AAA repair
3. Post endovascular stent grafting where stent stabilization is necessary due to stent fixation failure and/or persistent endoleak.

Exclusion Criteria:

1. Pregnant
2. Religious, cultural or other objection to the receipt of blood, or blood products.
3. Unwilling to comply with follow-up schedule
4. Unwillingness, or inability to provide informed consent to both trila and procedure
5. Ruptured Aneurysm
6. Area where staple is to be placed has significant loose thrombus associated with it
7. Acute or chronic aortic dissection or mycotoc aneurysm
8. Allergy to device materials
9. Allergy to or intolerance to use of contrast media or cannot be exposed to suitable remedial treatment such as steroids and/or diphenhydramine.
10. Clinically and morbidly obese such that imaging would be severely adversely affected.
11. Uncorrectable bleeding abnormality
12. Inflammatory aneurysm
13. Connective tissue disease (e.g., Marfans syndrome, Ehlers Danlos syndrome)
14. Patients with PTFE grafts
15. Patients with investigational grafts (i.e., those grafts that are not FDA approved)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Arko, MD, Study Chair — St. Paul University Hospital, Dallas Texas; Peter Faries, MD, Principal Investigator — Mount Sinai Hospital, New York; Louis Sanchez, MD, Principal Investigator — Barnes Jewish Hospital, St. Louis Missouri; Venkatash Ramaiah, MD, Principal Investigator — Arizona Heart Institute, Phoenix, Arizona; Mark Mewissen, MD, Principal Investigator — St. Luke's Medical Center; Mark Fillinger, MD, Principal Investigator — Mary Hitchcock Memorial Hospital, Lebanon New Hampshire; Zvonko Krajcer, MD, Principal Investigator — St. Lukes Episcopal Hospital, Houston Texas; Will Jordan, MD, Principal Investigator — University of Alabama, Birmingham Alabama.; Anthony Lee, MD, Principal Investigator — University of Florida, Gainesville, Florida; Karthikes Kasirajan, MD, Principal Investigator — Emory University, Atlanta Georgia
Locations (7):
- United States (7):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Arizona Heart Hospital, Phoenix, Arizona
  - Emory University Hospital, Atlanta, Georgia
  - Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - Mount Sinai Hospital, New York, New York
  - St. Paul University Hospital, Dallas, Texas
  - St. Lukes Episcopal Hospital, Houston, Texas